CLINICAL TRIAL: NCT07303803
Title: Chiglitazar in Combination With Anti-Inflammatory and Hepatoprotective Therapy for the Treatment in MASH Associated With T2DM: a Prospective, Multicentre, Randomised, Double-blind, Placebo-controlled Study
Brief Title: A Study of Chiglitazar in Patients With Metabolic Dysfunction-associated Steatohepatitis and Type 2 Diabetes Mellitus
Acronym: CHIG-MASH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Principal Investigator, Hai Li, Professor, Department of Gastroenterology, Punan Campus, RenJi Hospital, Shanghai Punan Hospital of Pudong New District
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KS2540
Record Dates: First submitted 2025-12-11; First posted 2025-12-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: MASH - Metabolic Dysfunction-Associated Steatohepatitis; T2DM (Type 2 Diabetes Mellitus)
Keywords: chiglitazar; metabolic dysfunction-associated steatohepatitis; type 2 diabetes; liver biopsy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — chiglitazar; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiglitazar Placebo + vitamin E + polyene phosphatidyl choline (Placebo Comparator): Chiglitazar placebo given orally once a day
  Interventions: Drug: Chiglitazar Placebo; Drug: vitamin E; Drug: Polyene Phosphatidyl choline
- 48mg Chiglitazar + vitamin E + polyene phosphatidyl choline (Experimental): 48mg Chiglitazar given orally once a day
  Interventions: Drug: Chiglitazar; Drug: vitamin E; Drug: Polyene Phosphatidyl choline

INTERVENTIONS:
Drug: Chiglitazar Placebo — Chiglitazar Placebo 48mg/day
  Other Names: simulant of chiglitazar
  Arms: Chiglitazar Placebo + vitamin E + polyene phosphatidyl choline
Drug: Chiglitazar — Chiglitazar 48mg/day
  Other Names: Carfloglitazar
  Arms: 48mg Chiglitazar + vitamin E + polyene phosphatidyl choline
Drug: vitamin E — Vitamin E 100mg/three times a day
  Other Names: Laiyi
Drug: Polyene Phosphatidyl choline — Polyene Phosphatidyl choline 456mg/three times a day
  Other Names: Yi Shan Fu

SUMMARY:
This trial aims to evaluate the efficacy and safety of chiglitazar as a combination therapy for patients with MASH and T2DM.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatohepatitis (MASH), used to be called non-alcoholic steatohepatitis (NASH), is a manifestation of the metabolic syndrome in the liver, particularly when co-occurring with type 2 diabetes (T2DM), presents a significant therapeutic challenge due to a higher risk of fibrosis progression and adverse outcomes. While new treatments for MASH are emerging, their efficacy in the T2DM subpopulation remains an area of unmet need. Chiglitazar is a novel peroxisome proliferator-activated receptor (PPAR) pan-agonist that regulates key pathways in lipid metabolism, glucose homeostasis, and inflammation. This trial aims to evaluate the efficacy and safety of chiglitazar as a combination therapy for patients with MASH and T2DM.

This is a prospective, multicentre, randomised, double-blind, placebo-controlled study. The trial will enroll 300 adult patients aged 18-75 years with biopsy-confirmed MASH and fibrosis stage F1 or higher. Participants will be randomised (1:1) to receive either chiglitazar 48 mg daily or a matching placebo. All participants will also receive background therapy consisting of vitamin E (100 mg three times a day) and polyene phosphatidylcholine (456 mg three times a day). The treatment duration is 78 weeks. The primary efficacy endpoint is the resolution of steatohepatitis with no worsening of liver fibrosis. Key secondary endpoints include improvement in liver fibrosis by at least one stage and changes in metabolic and liver safety biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged at least 18 years and under 75 years (inclusive) at the time of obtaining consent.
2. Participants must be diagnosed as T2DM and HbA1c ≤ 9.5% at time of screening.
3. Participants must take Fibroscan examination with the result of CAP ≥ 238 dB/m and LSM>8.5 kPa.
4. Diagnosis of MASH by liver biopsy, with NAFLD Activity Score (NAS) ≥4 with ≥1 point for each component, and fibrosis stage 1 or more over according to the NASH Clinical Research Network (CRN) scoring system. (or liver biopsy not more than 6 months prior to screening)
5. Stable body weight (≤10% body weight change) for at least 3 months.
6. Possess good understanding and behavior and be able to take the medication daily as required by the trial.
7. Willing to sign the informed consent.

Exclusion Criteria:

1. Alcohol consumption >20g ethyl alcohol/day for women and >40g ethyl alcohol/day for men.
2. Evidence of other forms of chronic liver disease:

   1. Alcoholic liver disease,
   2. Hepatitis B as defined by presence of hepatitis B surface antigen (HBsAg) or hepatitis B DNA,
   3. Hepatitis C as defined by presence of hepatitis C virus (HCV) RNA or positive hepatitis C antibody (anti-HCV),
   4. Evidence of autoimmune liver disease as defined by compatible liver histology,
   5. Current drug-induced liver disease as defined on the basis of typical exposure and history,
   6. Suspected or proven liver cancer,
   7. Any other type of liver disease other than MASH.
3. Uncontrolled T2DM defined as HbA1c >9.5% at time of screening or Type 1 diabetes mellitus (T1DM).
4. Patients with T2DM who have a history of diabetic ketoacidosis, proliferative diabetic retinopathy, diabetic maculopathy or severe non-proliferative diabetic retinopathy that requires acute treatment.
5. Any of the following cardiovascular conditions within 6 months prior to screening:

   1. acute myocardial infarction (MI),
   2. cerebrovascular accident (stroke),
   3. unstable angina,
   4. hospitalization due to congestive heart failure (CHF)
   5. New York Heart Association Functional Classification IV CHF
6. History of an active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
7. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg).
8. Renal impairment measured as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2.
9. Known clinically significant gastric emptying abnormality (for example, severe diabetic gastroparesis or gastric outlet obstruction) or chronically take drugs that directly affect gastrointestinal motility.
10. Have a known self or family history (first-degree relative) of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or medullary thyroid carcinoma (MTC).
11. Evidence of untreated hypothyroidism or hyperthyroidism based on clinical or laboratory evaluation.
12. A transplanted organ (corneal transplants allowed) or awaiting an organ transplant.
13. Women of childbearing potential: positive pregnancy test during screening or at randomization or unwillingness to use an effective form of birth control during the trial (at least include one barrier contraceptive method) and breast feeding.
14. Use of drugs associated with hepatic steatosis (e.g., amiodarone, methotrexate, tamoxifen) for more than 2 weeks in the 3 months prior to screening.
15. Current use of medication is associated with weight gain, except when on stable dose for at least 3 months prior to screening and remaining on stable dose during the study.
16. Receiving or having received (within 3 months of screening) chronic (>2 weeks) systemic glucocorticoid therapy.
17. Use of medications or alternative remedies (within 3 months prior to screening; prescribed or over-the-counter) intended to promote weight loss.
18. Use of treatment targeting MASH for more than 2 weeks in the 3 months prior to screening (GLP-1 receptor agonists, TZD analogues or PPAR pan agonists).
19. Any other condition which in the opinion of investigator would impede compliance or hinder completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with resolution of steatohepatitis and no worsening of liver fibrosis | week 78
  The definition of resolution of steatohepatitis was based on the following criteria: either a reduction in NAS score of at least 2 points or a post-treatment NAS score of 3 points or less; a minimum 1-point improvement in score for ballooning or inflammation

SECONDARY OUTCOMES:
Percentage of participants with an improvement in liver fibrosis by ≥ 1 stage (NASH CRN fibrosis score) and no worsening of steatohepatitis | week 78
  Evaluation of fibrosis stage was based on the nonalcoholic steatohepatitis clinical research network (NASH CRN) fibrosis staging system, participants were evaluated with the NASH CRN scoring system with ≥1-point reduction without worsening of MASH (defined as no increase in the NAS score).
Percentage of participants with resolution of steatohepatitis and improvement in liver fibrosis | week 78
  Participants were evaluated with the NASH CRN scoring system with ≥1-point reduction and with resolution of steatohepatitis
Change in body mass index from baseline | Week 2, 6, 13, 26, 39, 52, 65, 78
  The body mass index = weight (kg) / height (m)².
Changes in liver stiffness values assessed by transient elastography from baseline | Week 2, 6, 13, 26, 39, 52, 65, 78
  Measured by Fibroscan, to evlaute the severity of liver fibrosis
Change in CAP values assessed by transient elastography from baseline | Week 2, 6, 13, 26, 39, 52, 65, 78
  Measured by Fibroscan, to evlaute the severity of liver fat
Change in HbA1c from baseline | Week 2, 6, 13, 26, 39, 52, 65, 78
  Central lab test
Changes in blood fasting plasma glucose level from baseline | Week 2, 6, 13, 26, 39, 52, 65, 78
  Central lab test
Changes of blood lipids level from baseline | Week 2, 6, 13, 26, 39, 52, 65, 78
  Includeing TC, LDL-C, HDL-C, VLDL-C, non-HDL-C, TG
Changes of liver function from baseline | Week 2, 6, 13, 26, 39, 52, 65, 78
  Includeing AST, ALT, GGT, AKP

CONTACTS AND LOCATIONS:
Overall Officials: Hai Li, professor, Principal Investigator — Shanghai Punan Hospital of Pudong New District (Punan Branch of Renji Hospital, Shanghai Jiaotong University School of Medicine)
Locations (17):
- China (17):
  - Ditan Hospital of integrated traditional Chinese and Western Medicine Center, Beijing, Beijing Municipality
  - Southwest Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Southern Hospital, Guangzhou, Guangdong
  - Wuhan Union Hospital of Huazhong University of Science and Technology, Wuhan, Hebei
  - Taihe Hospital, Shiyan, Hubei
  - Xiangya hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Renji hospital of Shanghai Jiao Tong University School of Medical, Shanghai, Shanghai Municipality
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Shanghai Punan Hospital of Pudong New District (Punan Branch of Renji Hospital, Shanghai Jiaotong University School of Medicine), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No